CLINICAL TRIAL: NCT04702581
Title: A Randomized Trial of Delayed Radiotherapy in Patients 1p/19q Codeleted Low-grade Oligodendrogliomas Requiring a Treatment Other Than Surgery
Brief Title: A Randomized Trial of Delayed Radiotherapy in Patients Low-grade Oligodendrogliomas Requiring a Treatment Other Than Surgery
Acronym: POLO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0073; 2020-A02646-33 (Other: IDRCB)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Oligodendroglioma; Low-grade Oligodendroglioma; 1p19q Codeletion
Keywords: low-grade oligodendroglioma; radiotherapy; PCV; neurocognitive deterioration
MeSH Terms: conditions — Oligodendroglioma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCV alone (Experimental): Administration of 6 cycles of PCV chemotherapy alone.
  Interventions: Drug: PCV chemotherapy
- RT + PCV (Active Comparator): Radiotherapy followed by administration of PCV chemotherapy.
  Interventions: Drug: Radiotherapy and PCV chemotherapy

INTERVENTIONS:
Drug: PCV chemotherapy — 1. cycle of PCV chemotherapy is given as:
     * Day 1: CCNU 110 mg/m2 orally;
     * Days 8 and 29: Vincristine 1.4 mg/m2 IV;
     * Days 8 to 21: Procarbazine 60 mg/m2 orally
  6 cycles are given.
  Arms: PCV alone
Drug: Radiotherapy and PCV chemotherapy — Radiotherapy will deliver 50.4 Gy in 28 fractions of 1.8 Gy using IMRT technique.
  Followed by 6 cycles of PCV chemotherapy
  1 cycle of PCV is given as:
  * Day 1: CCNU 110 mg/m2 orally;
  * Days 8 and 29: Vincristine 1.4 mg/m2 IV;
  * Days 8 to 21: Procarbazine 60 mg/m2 orally
  Arms: RT + PCV

SUMMARY:
Because of their prolonged survival, patients with 1p/19q-codeleted low-grade oligodendrogliomas treated with RT + PCV are at risk of neurocognitive deterioration. We make the hypothesis that withholding radiotherapy until tumor progression could reduce the risk of neurocognitive deterioration without impairing overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Tumor is co-deleted for 1p and 19q based and IDH-mutant (IDH1 or IDH2) according to local diagnosis
* Histological confirmation of low-grade oligodendroglioma by central pathological review according to WHO 2016 classification
* Age ≥ 18 years
* Patients with one or several prior surgical procedure for a low-grade oligodendroglioma and who undergo a resurgery are eligible if they have not received prior radiotheray or chemotherapy and if the last histological diagnosis is a low-grade oligodendroglioma prior use of specific HDI prohibitions is permitted
* Patients who undergo an initial follow-up after surgery or re-surgery are eligible if there is no evidence of anaplastic transformation on MRI (no new contrast enhancement, no obvious modification of the growth rate)
* Patients requiring an oncological treatment other than surgery because of one or more of the following characteristics:

  * Progressive disease defined as documented growth prior to inclusion
  * Symptomatic disease defined as the presence of neurological or cognitive symptoms or refractory seizures defined as having both persistent seizures interfering with everyday life activities other than driving a car and three lines of anti-epileptic drug regimen had not worked, including at least one combination regimen.
  * Age ≥ 40 and any surgical therapy
  * Age < 40 with prior and subtotal resection or biopsy (i.e., anything less than gross total resection)
* Willing and able to complete neurocognitive examination and the QOL
* Karnofsky performance status ≥ 60
* Laboratory values obtained between 21 days before inclusion andrandomization, respecting the following criteria:
* Absolute neutrophil count (ANC) ≥1500 /mm3
* Platelet count ≥100,000 / mm3
* Hemoglobin > 9.0 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* SGOT (AST) ≤ 3 x ULN
* Negative serum or urine pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only.
* Provide informed written consent

Exclusion Criteria:

* Pregnant and nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception for up to 6 months following the completion of PCV.
* Received any prior radiation therapy or chemotherapy for any CNS neoplasm.
* Co-morbid systemic illnesses or other severe concurrent disease which would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Concomitant serious immunocompromised status (other than that related to concomitant steroids).
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm (except specific inhibitors of IDH)
* Other active malignancy within 5 years of registration. Exceptions: Non-melanotic skin cancer or carcinoma-in-situ of the cervix.
* Contra-indication to CCNU: hypersensitivity to CCNU, wheat allergy, association to yellow fever vaccin
* Contra-indication to Procarbazine: severe renal failure, severe hepatic failure, hypersensitivity to procarbazine, association to yellow fever vaccin
* Contra-indication to Vincristine: hypersensitivity to vincristine, neuromuscular disorder (for example demyelinating Charcot-Mary Tooth neuropathy), severe renal failure, severe hepatic failure.
* Not depending from the french system of health assurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival without neurocognitive deterioration | During 9 years
  Survival without neurocognitive deterioration (whatever the cause of deterioration, i.e toxicity or tumor progression) defined as the time from study randomization to failure in any of the 6 cognitive domains that will be explored (i.e memory, working memory, language, visuo-spatial ability, cognitive executive functions, behavioral executive functions) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression free survival | During 9 years
  Time from study randomization to the time of progression of the tumor
Overall survival | During 9 years
  Time from study randomization to the time of death

CONTACTS AND LOCATIONS:
Locations (26):
- France (26):
  - CHU d'Amiens-Picardie Site Sud, Amiens
  - Institut de Cancerologie de l'Ouest, Angers
  - CHU de Bordeaux Hôpital Saint André, Bordeaux
  - Institut de Cancérologie et Hematologie (ICH) - CHRU Brest, Hopital Morvan, Brest
  - Hospices Civils de Lyon, Bron
  - CHU de Caen, Caen
  - Hôpital d'Instruction des Armées PERCY, Clamart
  - Hôpital Pasteur - Hôpitaux civils de Colmar, Colmar
  - Centre Georges Francois Leclerc, Dijon
  - Hôpital Roger Salengro CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Timone, Marseille
  - CHU de Nice Hôpital Pasteur, Nice
  - Hôpital Saint-Louis, AP-HP, Paris
  - GH Pitié Salpêtrière, Paris
  - CH Annecy Genevois site Annecy, Pringy
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Centre de Lutte Contre le Cancer PAUL STRAUSS, Strasbourg
  - Hôpital Foch, Suresnes
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHRU de Tours, Tours
  - Gustave Roussy, Villejuif